CLINICAL TRIAL: NCT01775423
Title: A Phase I Clinical Study of BBI608 in Adult Patients With Advanced Malignancies
Brief Title: A Study of BBI608 in Adult Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-101
Record Dates: First submitted 2013-01-17; First posted 2013-01-25 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cancer, Advanced Malignancies
MeSH Terms: conditions — Neoplasms | interventions — napabucasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BBI608 (Experimental)
  Interventions: Drug: BBI608

INTERVENTIONS:
Drug: BBI608

SUMMARY:
This is an open label, single arm, dose escalation study of BBI608 in patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPPA) prior to study-specific screening procedures
2. For solid tumors or lymphoma, a histologically or cytologically confirmed solid tumor that is metastatic, unresectable, or recurrent and for which standard curative or palliative therapies do not exist or are no longer effective.
3. ≥ 18 years of age
4. For solid tumors, measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
5. For lymphoma, measurable disease as defined by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma
6. For multiple myeloma, measurable disease as defined by the International Uniform Response Criteria for Multiple Myeloma
7. Karnofsky performance status greater than or equal to 70%
8. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 dose
9. Females of childbearing potential must have a negative serum pregnancy test
10. Aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 1.5 × upper limit of normal(ULN)
11. Hemoglobin (Hgb) greater than or equal to 10 g/dl
12. Total bilirubin less than or equal to 1.5 × ULN
13. Creatinine less than or equal to 1.5 x ULN or creatinine clearance greater than 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal. Creatinine < 2.5 x ULN for multiple myeloma patients.
14. Absolute neutrophil count greater than or equal to 1.5 x 109/L
15. Platelets greater than or equal to 100 x 109/L
16. Life expectancy greater than or equal to 3 months

Exclusion Criteria

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of first dose with the exception for a single dose radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before beginning the administration of BBI608.
2. Surgery within 4 weeks prior to first dose
3. Any known untreated brain metastases. Treated subjects must be stable for 4 weeks after completion of that treatment, with image documentation required. Patients must have no clinical symptoms from brain metastases and must be either off steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated.
4. Pregnant or breastfeeding
5. Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection)
6. Unable or unwilling to swallow BBI608 capsules daily
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-03; Primary Completion 2015-08-06 (Actual); Study Completion 2015-08-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Adverse events will be assessed at baseline, while the participant is taking BBI608, and for 30 days after stopping therapy. The average length of this duration is expected to be approximately 4 months.
  Assessment of safety of BBI608 given in monotherapy to patients with advanced malignancies by reporting of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- Institute for Translational Oncology Research, Greenville Hospital System, Greenville, South Carolina, United States
- Canada (2):
  - Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec